CLINICAL TRIAL: NCT06887972
Title: A Phase 4, Open-label, Single-arm Study Evaluating the Effectiveness and Safety of Suzetrigine As Part of Multimodal Therapy for Acute Pain After Aesthetic or Reconstructive Surgeries
Brief Title: A Single-Arm Study Evaluating the Effectiveness and Safety of Suzetrigine (SUZ) for Acute Pain After Aesthetic or Reconstructive Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX24-548-113
Record Dates: First submitted 2025-03-19; First posted 2025-03-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Suzetrigine (SUZ) (Experimental): Participants will receive SUZ for 14 days or until their pain resolves, whichever occurs first.
  Interventions: Drug: Suzetrigine

INTERVENTIONS:
Drug: Suzetrigine — Tablets for oral administration.
  Other Names: VX-548; SUZ; JOURNAVX

SUMMARY:
The purpose of this study to evaluate the effectiveness, safety, and tolerability of SUZ as part of multimodal therapy (MMT) in treating acute postoperative pain.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of greater than or equal to (≥)18.0 to less than or equal to (≤) 40.0 kilogram per meter square (kg/m^2)
* Participants scheduled to undergo an aesthetic or reconstructive surgical procedure that would typically be treated with opioid therapy for at least 72 hours postoperatively

Key Exclusion Criteria:

• Participated in a previous study with SUZ or received Journavx

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants Reporting Good, Very Good, or Excellent on a Patient Global assessment (PGA) for Pain Control at the end of Treatment | From Day 3 up to Day 14

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center - Surgery, Boston, Massachusetts
  - HD Research LLC | First Surgical Hospital, Bellaire, Texas
  - Memorial Hermann Village, Houston, Texas
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/